CLINICAL TRIAL: NCT04227379
Title: Diabetes Disparities: Texting to Extend Treatment (DD-TXT)
Acronym: DD-TXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 17-087
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: text messaging; Health Equity; Health Care Quality, Access, and Evaluation; self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients who consented to participate were asked to complete the baseline survey instruments. Participants were then randomized to a study arm, using a separate randomization table per site. Since women are underrepresented among VHA patients, the study staff recruited women first to oversample them, with the goal of 10-20% women at each site. The goal was to recruit 400 participants (200 per site). Participants in both arms were asked to complete a follow-up survey and interview after completing the 6-month texting intervention they were assigned.
Who Masked: Participant
Masking Description: All participants received a diabetes self-management support texting intervention but they were not explicitly told whether their intervention was part of the experimental (DSMS+) or comparison (DSMS) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DSMS+ (DSMS Plus) (Experimental): Participants in this group were signed up for an interactive, patient-centered, and customizable diabetes self-management support texting intervention (DSMS+). This arm received the same daily educational content as the DSMS arm augmented by the following: regular two-way check-in messages about diabetes self-management behaviors, an invitation to receive messages written by other Veterans living with diabetes on demand, and a menu of optional and customizable modules (e.g., medication reminders, blood sugar and blood pressure monitoring,: physical activity reminders, weight management, and goal setting) from which participants could select messaging that supported their diabetes self-management goals. Patients could customize the timing and frequency of their messages. DSMS+ participants also received a once monthly message asking whether the messages had been helpful.
  Interventions: Behavioral: Intervention 1- DSMS+
- DSMS (Active Comparator): Participants in the comparison condition were signed up for a one-way education-only protocol called Diabetes Self-Management Support (DSMS), comprised of 6 months of once daily one-way text messages covering standard diabetes self-management education content. Starting with the VA educational workbook entitled "Self-Care Skills for the Person with Diabetes", created in alignment with VA/DoD diabetes guidelines, we enhanced the educational content by incorporating Veteran input through a co-design process with Veterans living with diabetes and expert clinician review. DSMS messages could not be customized. There was no interactive content for the DSMS arm other than a once monthly message asking whether the messages had been helpful.
  Interventions: Behavioral: Comparison - DSMS

INTERVENTIONS:
Behavioral: Intervention 1- DSMS+ — Participants in this group were signed up for an interactive, patient-centered, and customizable diabetes self-management support texting intervention (DSMS+). This arm received the same daily educational content as the DSMS arm augmented by the following: regular two-way check-in messages about diabetes self-management behaviors, an invitation to receive messages written by other Veterans living with diabetes on demand, and a menu of optional and customizable modules (e.g., medication reminders, blood sugar and blood pressure monitoring,: physical activity reminders, weight management, and goal setting) from which participants could select messaging th
  Other Names: DD-TXT
  Arms: DSMS+ (DSMS Plus)
Behavioral: Comparison - DSMS — Participants in the comparison condition were signed up for a one-way education-only protocol called Diabetes Self-Management Support (DSMS), comprised of 6 months of once daily one-way text messages covering standard diabetes self-management education content. Starting with the VA educational workbook entitled "Self-Care Skills for the Person with Diabetes", created in alignment with VA/DoD diabetes guidelines, we enhanced the educational content by incorporating Veteran input through a co-design process with Veterans living with diabetes and expert clinician review. DSMS messages could not be customized. There was no interactive content for the DSMS arm other than a once monthly message asking whether the messages had been helpful.
  Other Names: DSE
  Arms: DSMS

SUMMARY:
One way to help Veterans improve their diabetes control is through the use of technology to help provide information, motivation, and reminders necessary to support diabetes self-management. The study will seek input from diverse groups of Veterans living with diabetes to help develop a new customizable, interactive texting intervention that allows Veterans to choose what kinds of diabetes self-management support they need, and when. This diabetes support will be provided to Veterans through "Annie for Veterans", a VA texting system for self-management support. Patients will be randomized to receive a once-daily standard diabetes self-management texting intervention called DSMS based on standard diabetes self-management education content or a customizable, patient-centered diabetes self-management support intervention with additional features called DSMS Plus (DSMS+) in order to test the comparative effectiveness of these two texting interventions.

DETAILED DESCRIPTION:
Type 2 Diabetes is a common, complex health condition which can result in many serious and costly health complications if not treated and controlled properly. One in four Veterans are diagnosed with Type 2 Diabetes. Vulnerable Veterans, such as minority, low-income, or rural Veterans, and Veterans with comorbid mental health diagnoses, are disproportionately affected and are less likely to have their diabetes under control. The goal of this study, using a randomized comparative effectiveness design, was to test the comparative effectiveness of an interactive, customizable diabetes self-management support texting protocol (DSMS+), versus a standardized education-only intervention (DSMS) in a sample of Veterans with uncontrolled diabetes.

The team will invited Veterans age 18 years and above who were actively receiving care at the study sites (as determined by upcoming scheduled appointment) who had uncontrolled glucose (HbA1c >= 8.0% for at least 50% of the most recent 6 months). Participants who met these conditions and enrolled in the study were randomized to one of two study arms: DSMS or DSMS+. Both arms received text-based diabetes self-management support for 6 months. The primary outcome was HbA1c percent time in control. Secondary outcomes include self-reported adherence to diabetes self-care recommendations (SCI-R), diabetes self-efficacy, diabetes distress, LDL, and blood pressure control. The team hypothesized that the customizable texting intervention (DSMS+) would result in better proximal health outcomes and diabetes self-management behaviors vs a standardized, education-only protocol (DSMS).

Please note that we previously referred to DSMS as DSE (diabetes standardized education) and DSMS+ as DD-TXT (Diabetes Disparities: Texting to Extend Treatment) after the trial name. We updated the names to better clarify that both are diabetes self-management support texting interventions, with DSMS+ having additional, customizable and interactive content that patients can choose from.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Active VHA patients with type 2 diabetes
* Had at least 4 VA outpatient encounters in the previous year
* Have a future appointment scheduled, and not be hospitalized or institutionalized or have participated in Aim 1 DD-TXT development
* Have HbA1c lab data (2+ values) in the 12 months prior to RCT recruitment.
* Have inadequate glycemic control for at least 50% of the 6 months before invitation to participate.

Exclusion Criteria:

* Non-Veterans
* Not having access to their own or a cohabiting family member's cell phone or smartphone for participation
* Not willing and able to text
* A visual impairment that would prevent them from reading or replying to text messages
* Cognitively incapable of consent to participate (Failure of Short Blessed Test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
HbA1c percent time in control | 6 month follow up
  The investigators will examine the changes in HbA1c percent time in control. These data will be calculated using HbA1c measures pulled from the electronic medical record data.

SECONDARY OUTCOMES:
self-reported adherence to diabetes self-care recommendations (SCI-R) | 6 month follow up
  Secondary outcomes include self-reported adherence to diabetes self-care recommendations (SCI-R). These will be collected from the patient via a questionnaire conducted over the phone.
LDL | 6 month follow up
  Secondary outcomes include LDL. These data will be pulled from the electronic medical record data.
self-reported diabetes self-efficacy | 6 month follow up
  Secondary outcomes include self-reported adherence to diabetes self-efficacy. These will be collected from the patient via a questionnaire conducted over the phone.
self-reported diabetes distress | 6 month follow up
  Secondary outcomes include self-reported diabetes distress. These will be collected from the patient via a questionnaire conducted over the phone.
blood pressure control | 6 month follow up
  Secondary outcomes include blood pressure control. These data will be pulled from the electronic medical record data.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Shimada, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT04227379/ICF_000.pdf